CLINICAL TRIAL: NCT06592976
Title: Effects of Gut Microflora on Cervico-vaginal Microenvironment in Women with Endometriosis (Original Version: Effetti Della Flora Intestinale Sul Microambiente Cervico-vaginale in Donne Con Endometriosi)
Brief Title: Effects of a Multi-strain Oral Probiotic on the Vaginal Microbiota Composition in Healthy Women and Women with Endometriosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Marisa Di Pietro, Professor in Microbiology, University of Roma La Sapienza
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0751/2020
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Endometriosis; Bacterial Vaginosis; Healthy Volunteer
Keywords: Gut microbiota; Vaginal microbiota; Probiotic; endometriosis; bacterial vaginosis; 16s metagenomic
MeSH Terms: conditions — Endometriosis; Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Women with endometriosis (Experimental)
  Interventions: Dietary Supplement: Multi-strain Oral Probiotic (CDS22-formula)

INTERVENTIONS:
Dietary Supplement: Multi-strain Oral Probiotic (CDS22-formula) — All patients received the probiotic product CDS22-formula (also known under the tradenames Visbiome, De Simo-ne, Vivomixx) as acid-resistant oral capsules (twice daily for 2 months), containing 1.12 x 10^11 live bacteria per capsule.

SUMMARY:
Endometriosis is a chronic inflammatory disease affecting approximately 10-15% of reproductive age women, and, in recent years, an association between this pathology and dysbiosis, either involving the gut or the genital microbiota, has been hypothesized.

Therefore, the aim of the study is to investigate the etiopathogenetic role of cervico-vaginal microbiota, and its relationship to the gut microbiota, in women with endometriosis. Furthermore, the effects of a multi-strain oral probiotic formulation will be evaluated on the composition of the genital microbiota in healthy women and patients with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 40 years old;
* clinical diagnosis of endometriosis via gynecological examination and transvaginal ultrasound (TVUS);
* genital healthy condition as confirmed via gynecological examination.

Exclusion Criteria:

* pre-menarche or menopause status;
* diabetes, neoplastic diseases, urinary or genital infections in the past 6 months
* bowel and/or liver disorders;
* current treatment with oral contraceptive or progestins, prokinetics, antacids or proton pump in-hibitors;
* sexual activity in the week before sampling;
* recent or current antibiotic treatment (oral or topical);
* the use of probiotics and/or prebiotics for three months before the enrolment.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 123 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Comparison in the mean microbial diversity of the vaginal and gut microbiota between women with endometriosis and healthy volunteers, as assessed by Shannon Diversity Index (alpha-measure) and UniFrac analysis (beta measure), calculated in qiime2. | At the time of enrollment
  Microbial diversity through Shannon diversity index and UniFrac analysis will be calculated from the number and type of bacterial species in the vaginal and gut microbiota as assessed by the sequencing of the hypervariable region (v3-v4) of the bacterial 16s rDNA via metagenomic analysis (Illumina MiSeq platform).

SECONDARY OUTCOMES:
Changes in the mean microbial diversity (Shannon Diversity Index and UniFrac analysis) of the vaginal microbiota at two month supplementation, from baseline, of the probiotic product in either healthy women or women with endometriosis. | At the time of enrollment and after 2 months of probiotic supplementation
  Microbial diversity through Shannon diversity index (alpha measure) and UniFrac analysis (beta measure) will be calculated in qiime2 from the number and type of bacterial species in the vaginal and gut microbiota as assessed by the sequencing of the hypervariable region (v3-v4) of the bacterial 16s rDNA via metagenomic analysis (Illumina MiSeq platform).

CONTACTS AND LOCATIONS:
Locations (1):
- Umberto I Hospital, University of Rome "Sapienza", Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No